CLINICAL TRIAL: NCT03839563
Title: Temporal Relations and Exercise Interventions of Various Gait and Cognitive Domains in Older Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Medical University (Other)
Collaborators: National Health Research Institutes, Taiwan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NHRI-EX108-10804PI
Record Dates: First submitted 2019-01-31; First posted 2019-02-15 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Fallers; Mild Cognitive Impairment
Keywords: Biomarker; Cognitive impairment; Gait abnormality; Older Adults; Exercise
MeSH Terms: conditions — Cognitive Dysfunction; Mobility Limitation; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: A pragmatic, single-blinded, randomized controlled trial with three arms will be conducted to investigate the effectiveness of conventional exercise and tai chi chuan, compared to health education/usual physical activity.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional exercise (Experimental): This exercise will comprise stretching, muscle strengthening, and balance training at increasing difficulty levels, tailored and supervised by a physical therapist, and will take place at a subject's residence or in the neighborhood once a week for 6 months. Each session will last 60 min.
  Interventions: Behavioral: Exercise
- Tai chi chuan (Experimental): The 8-form Yang-style tai chi chuan intervention will take place at a subject's residence or in the neighborhood once a week for 6 months, and each session will last 60 min.
  Interventions: Behavioral: Exercise
- Health education/usual physical activity (No Intervention): After the baseline, the case manager will visit subjects in this group once for comparability with the other two intervention groups and instruct them to maintain their usual physical activity.

INTERVENTIONS:
Behavioral: Exercise — Each session will last 60 min, consisting of 10 min of warm-up, 45 min of exercise, and a 5-min cool-down.
  Arms: Conventional exercise; Tai chi chuan

SUMMARY:
The effectiveness of conventional exercise, tai chi chuan and health education/usual physical activity over a 6-month intervention period in improving primary outcomes and secondary outcomes in older mild cognitive impairment adults will be compared. Third, whether changes in serum levels of the brain-derived neurotrophic factor (BDNF), insulin-like growth factor (IGF)-1, and vascular endothelial growth factor (VEGF) and expression of the apolipoprotein E (APOE) ε4 allele parallel changes in gait characteristics and cognitive functions after the intervention will be examined.

ELIGIBILITY:
Inclusion Criteria:

* At least 65 years old
* Had an emergency department visit due to a fall at least 3 months prior to the baseline assessment (assuming a full recovery time from a fall to be 3 months)
* Can ambulate independently
* Has mild cognitive impairment

Exclusion Criteria:

* Do not live in a community setting
* Cannot ambulate independently and communicate with researchers
* Have a major unstable cardiopulmonary disease (e.g., ischemic chest pain, shortness of breath, recurrent syncopal episodes, orthopnea, paroxysmal nocturnal dyspnea, palpitations, or tachycardia)
* Have a contraindication to physical exercise (e.g., severe osteoarthritis or severe pulmonary hypertension)

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 189 (Estimated)
Dates: Start 2019-02-15 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Gait characteristics | 12 months
  Performance on six gait characteristics (velocity, cadence, stride length, swing time, stride length variability, and swing time variability) will be measured with a 6-m electronic walkway of GAITRite.
Global cognition | 12 months
  Global cognition will be assessed using the Mini-Mental State Examination (MMSE). The MMSE comprises 11 questions, and the score ranges 0~30, with lower scores indicating poorer global cognition.
Serum levels of BDNF | 12 months
  Serum BDNF concentrations will be assessed.
Serum levels of IGF-1 | 12 months
  Serum IGF-1 concentrations will be assessed.
Serum levels of VEGF | 12 months
  Serum VEGF concentrations will be assessed.

SECONDARY OUTCOMES:
Tinetti balance | 12 months
  The Tinetti balance score ranges 0~26, with a higher score indicating a better balance ability.
Mobility | 12 months
  The timed up and go test requires subjects to rise from a standard chair, walk a distance of 3 m, turn, walk back to the chair, and sit down. The time to complete the timed up and go will be recorded.
Muscle strength | 12 months
  Grip strength will be assessed via a handgrip dynamometer and measured in kilograms of isometric force.
Falls | 12 months
  number of falls and multiple falls
Depressive symptoms | 12 months
  Depressive symptoms will be assessed using the 15-item Geriatric Depression Scale (GDS).
Fear of falling | 12 months
  Fear of falling will be assessed using the Falls Efficacy Scale (FES) test.

CONTACTS AND LOCATIONS:
Overall Officials: Mau-Roung Lin, Professor, Principal Investigator — Taipei Medical University
Locations (1):
- Taipei Medical University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No